CLINICAL TRIAL: NCT05028309
Title: Effects of Obesity in the Aged
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tony Babb, PROFESSOR, Cardiopulmonary Laboratory Director, Effie and Wofford Cain Chair in Cardiopulmonary Research, Institute of Exercise and Environmental Medicine, Division of Pulmonary and Critical Care Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU-122010-108; 3R01AG070262-02S1 (NIH)
Record Dates: First submitted 2021-08-17; First posted 2021-08-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Aging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): Older group of adults (65-75 yrs). Everyone enrolled uses the 'intervention'/ external cuirass - mechanical unloading of thorax
  Interventions: Other: Mechanical unloading of the Thorax using an external cuirass

INTERVENTIONS:
Other: Mechanical unloading of the Thorax using an external cuirass — External cuirass (i.e., a plastic shell over the thorax) will be used to mechanically unload the chest wall. The cuirass has different operating modes. It can generate a constant negative pressure over the chest wall (e.g., -20cmH2O) or it can be triggered off mouth flow so it can generate a negative pressure on the chest wall during inspiration (e.g., -21cmH2O) and a positive pressure during expiration (e.g., +7cmH2O).

SUMMARY:
The overall objective of this application is to investigate the effects of obesity on lung function, exercise tolerance, and DOE in older obese adults as compared with older adults without obesity, using a novel probe for mechanically unloading the thorax at rest and during exercise. The investigators will use 1) continuous negative cuirass pressure, and 2) assisted biphasic cuirass ventilation to decrease obesity-related effects in older obese adults. Our approach will be to examine respiratory function, exercise tolerance, and DOE with and without mechanical unloading in older obese men and women (65-75 yr), including those with respiratory symptoms (defined by a score of 1 or 2 on the modified Medical Research Council Dyspnea Scale), as compared with older adults without obesity.

Specific Aims: The investigators will test the following hypotheses in older adults with and without obesity:

Aim 1) Obesity will decrease respiratory function but to a greater extent in older obese adults with respiratory symptoms, (as evidenced by altered pulmonary function and breathing mechanics at rest); Aim 2) Obesity will decrease exercise tolerance (as evidenced by peak V•O2 in ml/min/kg, i.e., physical fitness), but not cardiorespiratory fitness (as evidenced by peak V•O2 in % of predicted based on ideal body wt), except in older obese adults with respiratory symptoms where both may be reduced during graded cycle ergometry.

Aim 3) Obesity will increase DOE but to a greater extent in older obese adults with respiratory symptoms as evidenced by increased ratings of perceived breathlessness (sensory & affective dimensions) during exercise.

Aim 4) Mechanical unloading of the thorax will improve respiratory function, submaximal exercise tolerance, and DOE in older obese adults, but to a greater extent in older obese adults with respiratory symptoms.

DETAILED DESCRIPTION:
Over 40% of older adults (60+ yr) are obese and 30% are overweight. While regular exercise is an important component in the prevention and treatment of obesity, many older adults with obesity are unable or unwilling to exercise due to exercise intolerance and/or dyspnea on exertion (DOE). The Investigators have identified numerous obesity-related respiratory effects that could influence exercise tolerance and DOE in younger obese adults including decreased pulmonary function altered respiratory mechanics increased work of breathing and increased metabolic demands of exercise. The Investigators have also identified many age-related ventilatory constraints in older adults without obesity. However, it is unclear whether these obesity-related and aging-related effects combine to reduce exercise tolerance, impose DOE, or contribute to respiratory symptoms in older obese adults. Respiratory symptoms in older adults are often wrongly diagnosed as deconditioning and/or cardiopulmonary disease, placing older obese adults at risk of costly clinical testing, unnecessary treatment, and potentially a reluctance to exercise, which is counterproductive to weight loss (WL) and the preservation of functional capacity, thus further diminishing their quality of life. The respiratory effects of obesity are underappreciated and have not been carefully examined in older adults, especially older obese adults with "respiratory symptoms" who may experience even greater respiratory effects.

The Investigators propose that many of the obesity-related respiratory effects in older obese adults are the result of low lung volume breathing, i.e., a reduction in functional residual capacity (FRC) at rest (seated upright & supine), and end-expiratory lung volume (EELV) during exercise. The Investigators suggest that increased fat on the chest wall (i.e., abdomen & rib cage) produces low FRC and EELV levels, where breathing limitations like expiratory flow limitation and enhanced perception of dyspnea are more likely to occur. This is because older adults have an age-related decline in maximal expiratory flow at low lung volumes. As such, excess fat on the thorax appears to exert an unfavorable burden on the older obese adult, particularly during exercise. Our overall hypothesis is that respiratory limitations, exercise intolerance, DOE, and respiratory symptoms in older obese adults are due to mechanical loading of the thorax and low lung volume breathing coupled with the age-related decline in maximal expiratory flow. The Investigators propose to test this hypothesis with the use of an external cuirass (i.e., a plastic shell over the thorax) to mechanically unload the chest wall.

Although our laboratory has used modest WL in younger obese women to reduce the effects of obesity, the mechanisms by which WL (i.e., decreased fat over the entire body) decreases DOE remain unclear. This may be in part due to our single global assessment of DOE (i.e., sensory domain only & pre-post WL only), and/or that changes in DOE in the time domain are not in parallel with WL. To circumvent these limitations of WL, an external cuirass will be used to mechanically unload the chest wall (includes rib cage & abdomen) in older obese adults. This will effectively decrease the load on the chest wall thereby increasing FRC at rest and EELV during exercise (i.e., via continuous negative cuirass pressure), and potentially decreasing the work of breathing during exercise (i.e., via assisted biphasic cuirass ventilation). This novel and quantifiable probe will allow us to investigate the effects of obesity in older adults and their influence on lung function, exercise tolerance, and DOE (sensory & affective dimensions). The proposed mechanistic studies would lead to a better understanding of the mechanical effects of obesity in older adults, which could alter testing and treatment strategies for older obese adults, especially those with exercise intolerance, DOE, and respiratory symptoms.

The overall objective of this application is to investigate the effects of obesity on lung function, exercise tolerance, and DOE in older obese adults as compared with older adults without obesity, using a novel probe for mechanically unloading the thorax at rest and during exercise. The Investigators will use 1) continuous negative cuirass pressure, and 2) assisted biphasic cuirass ventilation to decrease obesity-related effects in older obese adults. Our approach will be to examine respiratory function, exercise tolerance, and DOE with and without mechanical unloading in older obese men and women (65-75 yr), including those with respiratory symptoms (defined by a score of 1 or 2 on the modified Medical Research Council Dyspnea Scale), as compared with older adults without obesity.

Specific Aims: The Investigators will test the following hypotheses in older adults with and without obesity:

Aim 1) Obesity will decrease respiratory function but to a greater extent in older obese adults with respiratory symptoms, (as evidenced by altered pulmonary function and breathing mechanics at rest); Aim 2) Obesity will decrease exercise tolerance (as evidenced by peak V•O2 in ml/min/kg, i.e., physical fitness), but not cardiorespiratory fitness (as evidenced by peak V•O2 in % of predicted based on ideal body wt), except in older obese adults with respiratory symptoms where both may be reduced during graded cycle ergometry.

Aim 3) Obesity will increase DOE but to a greater extent in older obese adults with respiratory symptoms as evidenced by increased ratings of perceived breathlessness (sensory & affective dimensions) during exercise.

Aim 4) Mechanical unloading of the thorax will improve respiratory function, submaximal exercise tolerance, and DOE in older obese adults, but to a greater extent in older obese adults with respiratory symptoms.

The investigators' long-term objective is to examine the effects of obesity in older obese adults and provide novel results that could clarify the mechanisms of respiratory limitations, exercise intolerance, DOE, and/or obesity-related respiratory symptoms in older obese adults. Thus, these results will have broad and immediate clinical impact on the care of older adults with obesity, especially those with exercise intolerance, DOE, and/or respiratory symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy older adults 65-75 years of age with normal lung function; men 30< %body fat ≤50 and women 35< %body fat ≤55; and ability to perform pulmonary and exercise test. Other inclusion criteria include the following:
* Nonsmokers who have no history of smoking
* No personal history of significant mental illness
* No weight loss dietary restrictions
* No current or past history of significant substance or alcohol abuse
* No history, evidence, or uncontrolled symptoms of heart disease
* No history of uncontrolled hypertension
* No current medications that may interfere with exercise capacity
* No recent history or indication of asthma
* No musculoskeletal abnormality that would preclude exercise
* No serious health conditions that would preclude study goals or participation in exercise (per PI & medical staff & preliminary or follow up testing; including significant other diseases, occult asthma, prior surgeries-especial lung or abdominal, or history of chemotherapy that could affect lung or heart function)
* Only postmenopausal women will be included.
* Women on hormone replacement therapy will be allowed to participate if the dosage remains similar during the entire protocol.

Exclusion Criteria:

* Volunteers with a mMRC score of 3 or 4 will be excluded due to likeliness of underlying disease.
* Individuals participating in regular vigorous conditioning exercise such as running, jogging, aerobics, cycling, or swimming more than three times per week will be excluded. However, if subjects have an exceedingly high exercise capacity (greater than 2 SD of predicted), they will be excluded.
* Maximal cycle ergometry test will be used to determine if further participation in testing is appropriate for the participant (e.g., normal exercise test, exclude presence of provokable ECG changes suggestive of heart disease, or dangerous arrhythmias or exercise induced hypertension or bronchoconstriction. If the participant develops an abnormal ECG or shows other signs of exercise intolerance or if signs of cardiovascular disease are noted during the exercise test, it will be terminated and the participant will be referred to their personal physician for further evaluation (see DMSP).
* Premenopausal women will be excluded.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Function: Lung Volumes | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  Pulmonary function is comprised of several physiological variables but this study will primarily measure Lung Volume: FRC (liters) and TLC (liters)
Change in Exercise Tolerance - Peak VO2 | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic).
  Exercise Tolerance is represented by several physiological variables but the primary variable is Maximal oxygen uptake (L/min and percent predicted)
Change in Dyspnea on Exertion | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic).
  Dyspnea on Exertion is represented using the Borg Scale which provides Ratings of Perceived Breathlessness (RPB) during constant load exercise cycling. The Borg Scale measures from 0-10, where 0 = no breathlessness and 10 = maximal breathlessness.
Changes in PANAS Questionnaire | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic).
  Positive and Negative Affect Schedule. This scale consists of a number of words that describe different feelings and emotions.
Modified Medical Research Council Dyspnea Scale (mMRC Dyspnea Scale) | Outcome measures will be assessed immediately after completion of mMRC questionnaire (during study visit 2)
  Investigate the qualities of respiratory sensations (e.g., "effort of breathing", "breathing heavy", "breathing shallow") during exercise before and after mechanical unloading of the chest wall
Dyspnoea-12 | Outcome measures will be assessed immediately after completion of Dyspnoea-12 questionnaire (during study visit 2)
  This questionnaire is designed to help us learn more about how their breathing is troubling them.
ASI | Outcome measures will be assessed immediately after completion of ASI questionnaire (during study visit 2)
  The Anxiety Sensitivity Index (ASI) is a 16 item scale containing items specifying different concerns someone could have regarding their anxiety.
HADS | Outcome measures will be assessed immediately after completion of HADS questionnaire (during study visit 2)
  HADS (Hospital Anxiety and Depression Scale) aims to measure symptoms of anxiety (HADS Anxiety) and depression (HADS Depression). HADS score: 0-7 = normal; 8-10 = mild; 11-14 = moderate; 15-21 = severe
SDS-MC | Outcome measures will be assessed immediately after completion of MC-SDS questionnaire (during study visit 2)
  The Marlowe-Crowne Social Desirability Scale (MC-SDS) is a 33-item self-report questionnaire that assesses whether or not respondents are concerned with social approval.
IPAQ | Outcome measures will be assessed immediately after completion of IPAQ questionnaire (during study visit 2)
  International Physical Activity Questionnaires (IPAQ) is a 27-item self-reported measure of physical activity
WSQ | Outcome measures will be assessed immediately after completion of WSQ questionnaire (during study visit 2)
  Workforce Sitting Questionnaire (WSQ) is to estimate how much time they usually spend sitting in each of the following activities on a working day and a non-working day.
SF-12 | Outcome measures will be assessed immediately after completion of SF-12 questionnaire (during study visit 2)
  SF-12 is a health-related quality-of-life questionnaire

SECONDARY OUTCOMES:
Changes in forced vital capacity (FVC) | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  FVC is the total amount of air (liters) exhaled during the forced expiratory volume (FEV) lung function test during spirometry.
Changes in forced expiratory volume (FEV) | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  FEV is the amount of air (liters) a person can exhale during a forced breath. The amount of air exhaled is measured during the a lung function test during spirometry.
Changes in forced expiratory volume in 1 second (FEV1) | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  FEV1 is the maximum amount of air (liters) that the a participant can forcibly expel during the first second following maximal inhalation. The FEV1 is measured during the a lung function test during spirometry.
Changes in FEV1/FVC Ratio | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  The FEV1/FVC (%) ratio is a calculation often used to determine the presence of obstructive or restrictive lung diseases such as chronic obstructive pulmonary disease (COPD).
Changes is peak flow | ChangesOutcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic) between conditions (visits 3-6) compared to baseline between cohorts
  Peak flow measurement is done with a peak flow meter. It measures the maximum (or peak) speed at which air (liters/sec) can be blown out of the lungs. This measurement provides a general idea of how narrow the lung airways are. It can also show how much the airways are changing over time if measured each day.
Pulmonary Function: Diffusing Capacity | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  Diffusing Capacity: Diffusing capacity of lung for carbon monoxide(DLco) (ml/mmHg/min)
Exercise Tolerance: Work Rate | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  Associated variables such as work rate (W)
Exercise Tolerance: Minute Ventilation | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  Associated variables such as pulmonary ventilation (L/min)
Exercise Tolerance: Operational Lung Volumes | Outcome measures will be assessed within 24-48hrs after completion of each study condition (baseline, control, continuous, and dynamic)
  Associated variables such as operational lung volumes (EELV and EILV as a % of TLC)

CONTACTS AND LOCATIONS:
Overall Officials: Tony G Babb, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine, UT Southwestern and Texas Health Resources, Dallas, Texas, United States